CLINICAL TRIAL: NCT02983669
Title: The Effects of Zataria Multiflora Boiss (Shirazi's Thyme) on Biochemical Markers and Imaging Studies of Patients With Nonalcoholic Fatty Liver Disease (NAFLD)
Brief Title: The Effects of Zataria Multiflora Boiss (Shirazi's Thyme) on Nonalcoholic Fatty Liver Disease
Acronym: ThymeLiv
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mesbah Shams, MD, Associate professor of Internal medicine and Endocrinology, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 94-7648
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Fatty Liver; Fatty Liver, Nonalcoholic
Keywords: Thymus Plant; Multiflotriol [Supplementary Concept]; Zataria multiflora; Complementary Therapies; Herbal Medicine; Medicine, traditional
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thyme (Experimental): Zataria multiflora Boiss powder capsule 350 mg twice daily for 3 months
  Interventions: Dietary Supplement: Thyme
- Placebo (Placebo Comparator): Wheat powder capsule 350 mg twice daily for 3 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Thyme — Thyme capsule 350 mg twice daily
  Other Names: Shirazi's Thyme
  Arms: Thyme
Other: Placebo — Placebo capsule 350 mg twice daily
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the effects and safety of a dietary supplement, Zataria multiflora Boiss (Shirazi's Thyme) in the treatment of non alcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
In a randomized double-blind placebo-controlled clinical trial Shirazi's Thyme is compared with placebo. Investigators select randomly 90 patients with NAFLD by inclusion criteria. Investigators measure anthropometric and laboratory parameters including fasting blood sugar, insulin, liver enzymes, lipid profile, and grade in sonography before intervention and 90 days later. Patients are divided into two equal groups. Intervention group in addition to diet and exercise recommendations receive capsules containing 700 mg of Shirazi thyme powder daily for 90 days. Placebo group in addition to the same recommendations for diet and exercise, receives placebo capsules twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-65 years
* Body mass index: 18-35 kg/m2
* Serum ALT level: >45 U/Lit. in Males, >29 U/Lit. in Females
* Grade >=1 fatty liver in liver sonography

Exclusion Criteria:

* Pregnancy and Lactation
* Acute or chronic liver failure
* Acute or chronic renal failure
* Autoimmune or viral hepatitis
* Wilson's disease
* Diabetes mellitus
* Alcoholism
* Malignancy
* Hypothyroidism or hyperthyroidism
* Drug used in last three months: OCP, metformin, vitamin E, ursodeoxycholic acid, glucocorticoids, thiazolidenediones.
* History of allergic reactions to Thyme

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Change in ALT (Alanin aminotransferase) level | 3 months
Change in grade of fatty liver in sonography by use of Saverymuttu Scoring System | 3 months

SECONDARY OUTCOMES:
Change in AST (Aspartate aminotransferase) level | 3 months
Fasting blood sugar (FBS) | 3 months
Change in Gama GT (γ-glutamyl transpeptidase) level | 3 monyhs
Fasting insulin level | 3 months
Body weight | 3 months
Waist circumference | 3 months
Hip circumference | 3 months
Number of patients with adverse events | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Majid Nimruzi, MD, Principal Investigator — Research Center for Traditional Medicine & History of Medicine, Shiraz University of Medical Sciences, Shiraz, Iran; Mojtaba Heydari, MD, Principal Investigator — Research Center for Traditional Medicine & History of Medicine, Shiraz University of Medical Sciences, Shiraz, Iran; Nasrin dokht Zamani, MD, Principal Investigator — Research Center for Traditional Medicine & History of Medicine, Shiraz University of Medical Sciences, Shiraz, Iran
Locations (1):
- Shahid Motahhari Clinic, Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: Undecided